CLINICAL TRIAL: NCT04611035
Title: Q-GAIN (Using Qpop to Predict Treatment for GAstroIntestinal caNcer)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/00924
Record Dates: First submitted 2020-08-26; First posted 2020-11-02 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Gastrointestinal Cancer
Keywords: Qpop
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1.1 Tumour biopsies
  * maximum of 2 time points - baseline upon study enrolment and upon disease progression. Whenever possible, the tumour core biopsies will be performed under image guidance.
  * Up to 6 fresh core samples (each of Tumour and matched Adjacent-Normal/Non-Tumour) will be biopsied from each patient at each time-point.
  1.2 Blood -A total of 50ml or 3.5 tablespoons of blood will be taken during screening of the study. A total of 40mls or 2.5 tablespoons of blood will be taken prior to each chemotherapy cycle. At the end of study, a total of 40mls or 2.5 tablespoons of blood will be collected. In total, a maximum of about 330ml or 22 tablespoons of blood will be taken during the course of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patient with first-line gastrointestinal cancers and patient with advanced and refractory GI cancers (>1 line of treatment), or post-progression biopsy)
  Interventions: Device: QPOP

INTERVENTIONS:
Device: QPOP — QPOP will then be applied to establish the most efficacious drug combination for the specific organoid. Additional drugs other than those listed above may be screened depending on availability of cancer organoids. When patients progress after first-line treatment, QPOP generated second-line options will be informed to treating physicians and the physician will exercise his/her discretion to select the most suitable drug based on patient's comorbidities and organ function after a formal molecular/phenotype tumour board.

SUMMARY:
This is a multi-cohort proof of concept study involving patients with metastatic gastrointestinal cancers. In the first cohort of treatment-naïve patients, the investigators intend to create cancer organoids for 100 subjects. Then, the investigators intend to evaluate ex-vivo prediction of treatment outcomes using QPOP (see section 4.0 for detailed sample size calculation).

Patients enrolled on study will undergo a fresh biopsy of tumour lesion to obtain cells that will be used to generate patient-derived tumour organoids. These patients will go on to receive standard of care first-line chemotherapy +/- targeted therapy. Organoids will then be subjected to up to a 14-drug panel screening. The drugs in the respective drug panel have been shown to have activity in the respective cancers and would be used in the standard-of-care setting by treating physicians.

DETAILED DESCRIPTION:
Hypothesis: Ex-vivo sensitivity testing on patient derived tumour organoids using QPOP can identify drug combinations which may have clinical efficacy against metastatic gastrointestinal cancer.

Specific aim 1: To grow patients' gastrointestinal tumour-derived organoids.

Specific aim 2: To perform ex-vivo drug sensitivity testing on patient derived tumour organoids using QPOP for metastatic gastrointestinal cancers.

Specific aim 3: Asses the efficacy of phenotype directed therapy using QPOP to assign treatment after progression of standard of chemo for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

-

Patients may be included in the study only if they meet the following criteria:

1. Treatment naïve patient with gastrointestinal cancers (i.e. oesophageal, gastro-oesophgeal, gastric, small bowel, colorectal, hepatocellular, pancreatic and biliary tract) fit and planned for first line treatment, OR
2. Chemo-refractory patients with GI cancers deemed by investigator to be fit for clinical trial
3. Age ≥ 21 years
4. ECOG PS 0-1
5. At least 1 tumour lesion amenable to fresh biopsy
6. At least 1 measurable tumour lesion based on RECIST v 1.1 criteria
7. Estimated life expectancy of at least 24 weeks
8. Adequate organ function , including:

   1. Pre-biopsy

      o Bone marrow:
      * Absolute neutrophil (segmented and bands) count (ANC) ≥1.5 x 109/L
      * Platelets ≥ 100 x 109/L
      * Pro-Thrombin within ULN
      * Hemoglobin ≥ 8 x 109/L
   2. Pre-treatment

      * Bone marrow:

        * Absolute neutrophil (segmented and bands) count (ANC) ≥1.5 x 109/L
        * Platelets ≥ 100 x 109/L
        * Hemoglobin ≥ 8 x 109/L
      * Hepatic:

        * Bilirubin ≤ 1.5 x upper limit of normal (ULN),
        * ALT or AST ≤ 2.5x ULN, (or ≤ 5 X with liver metastases)
      * Renal:

        * Creatinine ≤ 1.5x ULN
9. Signed informed consent from patient or legal representative
10. Able to comply with study-related procedures.
11. Recovery from prior toxicity to G1, excluding alopecia.

Exclusion Criteria:

* There are no specific exclusion criteria if patients meet the inclusion criteria

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 20 patients with gastric cancer, and 80 patients with other GI cancers will be first be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Rates of radiological response | 3 years
  complete and partial clinical response, including confidence intervals.
Percentage of patients with successful organoid generation for each different tumour type. | 3 years
  Patients enrolled on study will undergo a fresh biopsy of tumour lesion to obtain cells that will be used to generate patient-derived tumour organoids.
Efficacy of second-line therapy | 3 years
  measured by Overall Response Rate for patients with gastric cancer.

SECONDARY OUTCOMES:
Haematologic and non-haematologic toxicities | 3 years
  Toxicity rating using the NCI CTC v4.03 scale

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cancer Genome Atlas Network. Comprehensive molecular characterization of human colon and rectal cancer. Nature. 2012 Jul 18;487(7407):330-7. doi: 10.1038/nature11252. PMID 22810696
- [Result] AACR Project GENIE Consortium. AACR Project GENIE: Powering Precision Medicine through an International Consortium. Cancer Discov. 2017 Aug;7(8):818-831. doi: 10.1158/2159-8290.CD-17-0151. Epub 2017 Jun 1. PMID 28572459